CLINICAL TRIAL: NCT03850834
Title: A Multiple-dose Study to Evaluate the Tolerability and Pharmacokinetics of Ammoxetine Hydrochloride Enteric-coated Tablets in Chinese Healthy Subjects
Brief Title: Study of Ammoxetine Hydrochloride Enteric-coated Tablets in Healthy Subject
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMXT201802/PRO
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ammoxetine Hydrochloride Enteric-coated Tablets (Experimental)
  Interventions: Drug: Ammoxetine Hydrochloride Enteric-coated Tablets
- Placebo Enteric-coated Tablets (Placebo Comparator)
  Interventions: Drug: placebo enteric-coated tablets

INTERVENTIONS:
Drug: Ammoxetine Hydrochloride Enteric-coated Tablets — There will be 3 ascending cohorts. The cohorts will be administered 15, 30, 45 mg q12h for 15 times. The results of each dose group were shown to be safe and tolerable, and then the next dose group was tested
  Arms: Ammoxetine Hydrochloride Enteric-coated Tablets
Drug: placebo enteric-coated tablets — There will be 3 ascending cohorts. The cohorts will be administered 15, 30, 45 mg q12h for 15 times. The results of each dose group were shown to be safe and tolerable, and then the next dose group was tested
  Arms: Placebo Enteric-coated Tablets

SUMMARY:
This study evaluates the safety, tolerability and pharmacokinetics of Ammoxetine Hydrochloride Enteric-coated Tablets in Chinese healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18-45 years
* Body weight ≥ 45kg (female) or 50Kg (male), 18 ≤ BMI ≤ 26
* Vital signs, physical examinations and laboratory tests and other tests prove participants are healthy
* Sign the informed consent form voluntarily and cooperate voluntarily to complete the test

Exclusion Criteria:

* Allergens (allergic to 2 or more drugs, food or pollen)
* comorbid illness (mental illness, liver and kidney disease, gastrointestinal diseases, nervous system disease, or other systemic diseases)
* have Clinically significant abnormal screening laboratory values.
* Systolic pressure > 140mmHg or diastolic > 90 mmHg
* Postural hypotension (systolic blood pressure drop by 20mmHg or diastolic blood pressure drop by 10mmHg after standing position)
* The QTc period ≥ 450ms (male) or 470ms (female) or has a history of QTc extension
* Smoking or alcohol consumption (14 units per week in the previous 4 weeks : 1 unit = beer 285mL, or 25mL of spirits, or 150 mL of wine; Daily smoking ≥ 5) or abusing in past year of drug and other substance
* Have donated or lost blood 400 ml within 8 weeks prior to screening
* Participated in other clinical trials within 3 months prior to screening
* Intakes too much caffeinated beverage or food within 4 weeks prior to screening. such as: Coffee, tea, chocolate, cola, red bull (no more than 6 units per day). 1 unit of caffeine = 1 cup of coffee (177.4 mL) = 2 pots of cola (354.9 mL) = 1 cup of tea (354.9 mL) = 1/2 cup energy drink = 85g chocolate
* Have taken drugs that changed liver enzyme activity, such as dexamethasone, ketoconazole, rifampicin and omeprazole, were used within 4 weeks prior to screening
* Have taken prescription drugs and OTC (except for the occasional use of acetaminophen and nasal sprays), herbs vitamins or minerals within 4 weeks prior to screening. The interval from prior treatment to screening should be at least 5 half-lives metablism which subjected to the longer halflife
* Using any psychotropic drug or psychoactive substance
* Women were screened for positive blood pregnancy
* The subjects and their partners were not willing to take contraceptives during trial and six months after the study
* Have a donor plan recently
* Have participated in this trial
* The researchers believe that anyone who is unfit to participate in this test will be involved

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-03-10 (Estimated); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Event | 15 days
  Incidence of Adverse Events that researchers determined clinical significance
Area under the plasma concentration time curve (AUC) | 11 days
  The pharmacokinetics(PK) profile of Ammoxetine Hydrochloride Enteric-coated Tablets
Maximum concentration (Cmax) | 11 days
  The pharmacokinetics(PK) profile of Ammoxetine Hydrochloride Enteric-coated Tablets
Half life Period (t1/2) | 11 days
  The pharmacokinetics(PK) profile of Ammoxetine Hydrochloride Enteric-coated Tablets